CLINICAL TRIAL: NCT02971254
Title: The Effects of Inhalational Anaesthetics in Cognitive Functions in Down Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Gkliatis Emmanouil, Anaesthetist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8174
Record Dates: First submitted 2016-11-11; First posted 2016-11-22 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Down Syndrome
Keywords: cognitive functions; anaesthesia recovery; sevoflurane; desflurane
MeSH Terms: conditions — Down Syndrome | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane group (Active Comparator): inhalation anaesthetic Sevoflurane, 1 M.A.C. during surgery
  Interventions: Drug: Sevoflurane
- Desflurane group (Active Comparator): inhalation anaesthetic Desflurane, 1 M.A.C. during surgery
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Sevoflurane group
Drug: Desflurane
  Arms: Desflurane group

SUMMARY:
Recovery of the cognitive functions and recovery features after general anaesthesia in Down syndrome patients. A comparison of Sevoflurane and Desflurane.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I, II or III
* Down syndrome patients
* must be able to undergone general anaesthesia
* dental surgery necessity

Exclusion Criteria:

* severe dementia
* severe hearing, vision, speaking problems

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Functions | Baseline (12 to 24 hours before surgery), 1,5 hours after surgery and 4 hours after surgery
  Quantitative result measured by Prudhoe Cognitive Function Test (PCFT), a scale to assess cognitive function in adults with Down's syndrome.

SECONDARY OUTCOMES:
Spontaneous breathing | Interval between discontinuation of inhaled agent and first spontaneous breath and up to 1 hour.
Eye opening | Interval between discontinuation of inhaled agent and first eye opening and up to 1 hour.
Extubation | Interval between discontinuation of inhaled agent and extubation and up to 1 hour.
Orientation | Interval between discontinuation of inhaled agent and orientation in place, time, people and up to 1 hour.
Respond to commands | Interval between discontinuation of inhaled agent and respond to commands and up to 1 hour.
modified Aldrete Scoring System (mASS) | Interval between entrance in Post Operative Care Unit (PACU) and fulfillment of the criteria mASS to discharge PACU and up to 2 hours.
Orientation in PACU | 30 minutes after PACU entrance
  Orientation in place, time and people in Post Operative Care Unit (PACU).
Orientation in PACU | 60 minutes after PACU entrance
  Orientation in place, time and people in Post Operative Care Unit (PACU).
Antiemetics necessity. | Interval between entrance in PACU and administer antiemetic medication and up to 4 hours.
  Note if additional antiemetics was needed up to 4 hours postoperatively.
Painkillers necessity. | Interval between entrance in PACU and administration of antiemetic medication and up to 4 hours.
  Note if additional painkillers was needed up to 4 hours postoperatively.
Patient Alertness, Wellness, Energy | Baseline, 12 to 24 hours before surgery
  Assessment of the accompanying persons.
Patient Alertness, Wellness, Energy | 1,5 hours after surgery
  Assessment of the accompanying persons.
Patient Alertness, Wellness, Energy | 4 hours after surgery
  Assessment of the accompanying persons.
Patient satisfaction over anaesthesia. | 4 hours after surgery
  Assessment of the accompanying persons.
Postanesthesia Discharge Scoring System (PADSS) | Fulfillment of the criteria of PADSS from discontinuation of inhaled agent and up to 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Gkliatis, MD, Principal Investigator — GH Asklepieio Voulas
Locations (1):
- Gkliatis Emmanouil, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gkliatis E, Makris A, Staikou C. The impact of inhalation anesthetics on early postoperative cognitive function and recovery characteristics in Down syndrome patients: a randomized, double - blind study. BMC Anesthesiol. 2021 Sep 17;21(1):227. doi: 10.1186/s12871-021-01447-x. PMID 34535086